CLINICAL TRIAL: NCT00041067
Title: Docetaxel (NSC-628503) And Vinorelbine (NSC-608210) Plus Filgrastim (NSC-614629) With Weekly Trastuzumab (NSC-688097) For HER-2 Positive, Stage IV Breast Cancer
Brief Title: S0215 Trastuzumab, Docetaxel, Vinorelbine, and Filgrastim in Treating Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069440; S0215 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Trastuzumab; Docetaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trastuzumab, docetaxel, vinorelbine and filgrastim (Experimental): Trastuzumab, docetaxel, vinorelbine and filgrastim
  Interventions: Biological: filgrastim; Biological: trastuzumab; Drug: docetaxel; Drug: vinorelbine

INTERVENTIONS:
Biological: filgrastim
Biological: trastuzumab
Drug: docetaxel
Drug: vinorelbine

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Colony-stimulating factors, such as filgrastim, may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combining trastuzumab with docetaxel, vinorelbine, and filgrastim in treating women who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 1-year survival of women with HER2-positive stage IV breast cancer treated with trastuzumab (Herceptin), docetaxel, and vinorelbine with filgrastim (G-CSF) support.
* Determine the response rate (complete and partial, confirmed and unconfirmed) in the subset of patients with measurable disease treated with this regimen.
* Determine the progression-free survival of patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Obtain tissue blocks for the determination of predictors of response (e.g., beta-tubulin mutations) to microtubule interacting agents in this patient population and for other future studies.

OUTLINE: This is a pilot, multicenter study.

Patients receive docetaxel IV over 1 hour on day 1, filgrastim (G-CSF) subcutaneously on days 2-21, vinorelbine IV over 6-10 minutes on days 8 and 15, and trastuzumab (Herceptin) IV over 30-90 minutes on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. If docetaxel and vinorelbine are discontinued due to unacceptable toxicity, patients may continue to receive trastuzumab. If trastuzumab is discontinued due to unacceptable toxicity, patients may continue to receive chemotherapy with G-CSF support.

Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 90 patients will be accrued for this study within 18-22.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV breast cancer

  * Metastasis to the ipsilateral supraclavicular lymph nodes allowed
* HER2-positive by fluorescence in situ hybridization (FISH) or immunohistochemistry 3+ staining confirmed in the adjuvant or metastatic setting
* No effusions or ascites as only sites of disease
* No primary or metastatic brain or central nervous system tumor
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin normal
* aspartate aminotransferase or Alanine aminotranferease no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN

Renal:

* Not specified

Cardiovascular:

* left ventricular ejection fraction normal by multigated radionuclide angiography or echocardiogram (patients who have received prior anthracycline therapy)
* No clinical evidence or history of cardiomyopathy

Other:

* No pre-existing grade 2 or greater motor or sensory peripheral neuropathy except abnormalities due to cancer
* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with Polysorbate 80
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other adequately treated stage I or II cancer currently in complete remission
* No known sensitivity to E. coli-derived proteins
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 months since prior chemotherapy
* Prior anthracycline as adjuvant therapy allowed
* No prior cumulative dose of doxorubicin more than 360 mg/m^2
* No prior cumulative dose of epirubicin more than 720 mg/m^2
* No more than 1 prior adjuvant or neoadjuvant chemotherapy regimen for primary disease
* No prior docetaxel
* No prior vinorelbine
* Prior paclitaxel allowed

Endocrine therapy:

* Prior hormonal therapy as adjuvant therapy or for metastatic breast cancer allowed
* No concurrent hormonal therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* At least 2 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2002-09; Primary Completion 2008-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Kash, MD, Study Chair — Edward Hospital Cancer Center
Locations (145):
- United States (145):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Ben E. Owens Cancer Treatment Center at St. Bernard's Medical Center, Jonesboro, Arkansas
  - Eden Medical Center, Castro Valley, California
  - Saint Rose Hospital, Hayward, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Lovelace Medical Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital Regional Cancer Center, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Livingston RB, Barlow WE, Kash JJ, Albain KS, Gralow JR, Lew DL, Flaherty LE, Royce ME, Hortobagyi GN. SWOG S0215: a phase II study of docetaxel and vinorelbine plus filgrastim with weekly trastuzumab for HER2-positive, stage IV breast cancer. Breast Cancer Res Treat. 2011 Nov;130(1):123-31. doi: 10.1007/s10549-011-1698-5. Epub 2011 Aug 9. PMID 21826527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the period February 2003 to December 2006, 76 patients were enrolled at 28 SWOG institutions.
Groups:
- Trastuzumab, Docetaxel, Vinorelbine and Filgrastim: Trastuzumab, docetaxel, vinorelbine and filgrastim
  docetaxel : 60 mg/m^2 on Day 1 of 21-day cycles
  vinorelbine : 27.5 mg/m^2 on Days 8 and 15
  filgrastim : 5 microg/kg/day on Days 2 to 21
  trastuzumab : 4 mg/kg by IV over a 90-minute period on Day 1 of the first cycle, then weekly 2 mg/kg by IV over a 30-minute period
Period: Overall Study
Arm/Group | Trastuzumab, Docetaxel, Vinorelbine and Filgrastim
Started | 76
Eligible | 74
Completed | 0
Not Completed | 76
Not completed — Adverse Event | 20
Not completed — Progression | 19
Not completed — Patient refusal | 12
Not completed — Other reasons | 23
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Trastuzumab, Docetaxel, Vinorelbine and Filgrastim
Number analyzed (Participants) | 74
Age, Customized [Number; unit: participants]
  30-39 | 11
  40-49 | 26
  50-59 | 19
  60-69 | 15
  70-79 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Survival at 1 Year
Time Frame: 1 year
Population: All eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Trastuzumab, Docetaxel, Vinorelbine and Filgrastim
Number analyzed (Participants) | 74
percentage of patients | 93 [84 to 97]

2. Secondary Outcome: Response Rate (Complete and Partial, Confirmed and Unconfirmed)
Description: Response was measured by the RECIST criteria. A patient was considered a responder if there was confirmed or unconfirmed partial or complete response. All others were considered non-responders even if the patient was technically not assessable due to different measurement techniques at the two time points.
Time Frame: response assessed after every 3 cycles (9 weeks) during treatment for up to 3 years if no progession
Population: patients with Response Evaluation Criteria in Solid Tumors measurable disease
Measure: Number; unit: participants
Arm/Group | Trastuzumab, Docetaxel, Vinorelbine and Filgrastim
Number analyzed (Participants) | 63
participants | 53 [63 to 84]

3. Secondary Outcome: Progression-free Survival
Time Frame: 2 years
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab, Docetaxel, Vinorelbine and Filgrastim
Number analyzed (Participants) | 74
months | 20 [15 to 28]

4. Secondary Outcome: Toxicity
Description: Number of patients for whom highest grade of toxicity observed during treatment. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: toxicities assessed every 3 weeks during treatment, for up to 3 years if no progession
Population: Eligible patients
Measure: Number; unit: Participants
Arm/Group | Docetaxel + Vinorelbine + G-CSF + Trastuzumab
Number analyzed (Participants) | 73
Participants
  Alkaline phosphatase increase | 1
  Anemia | 7
  Arthralgia | 1
  Bone pain | 2
  Catheter related infection | 2
  Chest pain,not cardio or pleur | 2
  Dehydration | 1
  Depression | 1
  Diarrhea without colostomy | 2
  Dyspepsia/heartburn | 1
  Dyspnea | 2
  Fatigue/malaise/lethargy | 9
  Febrile neutropenia | 4
  Headache | 3
  Hyperglycemia | 6
  Hypermagnesemia | 1
  Hypokalemia | 2
  Hypophosphatemia | 1
  Hypotension | 1
  Hypoxia | 1
  Infection w/o 3-4 neutropenia | 4
  Infection with 3-4 neutropenia | 1
  LVEF decrease/CHF | 1
  Leukopenia | 11
  Lymphopenia | 2
  Muscle weakness (not neuro) | 1
  Nausea | 3
  Neutropenia/granulocytopenia | 16
  PRBC transfusion | 1
  Pain-other | 3
  Pericar. effusion/pericarditis | 1
  Pneumonitis/infiltrates | 3
  Respiratory infect w/ neutrop | 1
  Respiratory infection, unk ANC | 1
  SGPT (ALT) increase | 1
  Sensory neuropathy | 5
  Syncope | 1
  Tearing | 1
  Thrombosis/embolism | 1
  Transplant-pRBC transfusion | 1
  Vomiting | 2

ADVERSE EVENTS:
Time Frame: Every 3 weeks for up to 3 years.
Description: Of the 74 eligible patients analyzed, one patient did not have toxicity assessments performed so only 73 patients are included in the adverse event evaluation.
Arm/Group | Docetaxel + Vinorelbine + G-CSF + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/73
Other Adverse Events (participants affected / at risk) | 71/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel + Vinorelbine + G-CSF + Trastuzumab (N=73)
Anemia (Blood and lymphatic system disorders) | 59
Febrile neutropenia (Blood and lymphatic system disorders) | 4
LVEF decrease/CHF (Cardiac disorders) | 4
Conjunctivitis (Eye disorders) | 5
Eye-other (Eye disorders) | 4
Tearing (Eye disorders) | 15
Abdominal pain/cramping (Gastrointestinal disorders) | 4
Constipation/bowel obstruction (Gastrointestinal disorders) | 16
Diarrhea without colostomy (Gastrointestinal disorders) | 32
Dyspepsia/heartburn (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 26
Stomatitis/pharyngitis (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 12
Edema (General disorders) | 18
Fatigue/malaise/lethargy (General disorders) | 63
Fever without neutropenia (General disorders) | 11
Pain-other (General disorders) | 15
Rigors/chills (General disorders) | 5
Infection w/o 3-4 neutropenia (Infections and infestations) | 12
Alkaline phosphatase increase (Investigations) | 40
Bilirubin increase (Investigations) | 4
Leukopenia (Investigations) | 23
Neutropenia/granulocytopenia (Investigations) | 24
SGOT (AST) increase (Investigations) | 17
SGPT (ALT) increase (Investigations) | 14
Thrombocytopenia (Investigations) | 9
Weight loss (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 5
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 33
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 5
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 24
Dizziness/light headedness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 15
Neuropathic pain (Nervous system disorders) | 5
Sensory neuropathy (Nervous system disorders) | 35
Taste disturbance (Nervous system disorders) | 12
Anxiety/agitation (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 16
Dysuria (Renal and urinary disorders) | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 43
Nail changes (Skin and subcutaneous tissue disorders) | 16
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Hot flashes (Vascular disorders) | 6
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No